CLINICAL TRIAL: NCT04512339
Title: Dupilumab in Severe Chronic Hand Eczema With Inadequate Response or Intolerance to Alitretinoin
Brief Title: Dupilumab in Severe Chronic Hand Eczema
Acronym: DUPSHE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Marie Louise A Schuttelaar, MD, PhD, Principal Investigator, Dermatologist, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201900237
Record Dates: First submitted 2020-06-12; First posted 2020-08-13 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hand Eczema
Keywords: Hand eczema; Dupilumab
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: 2:1 randomization. Two-thirds will receive dupilumab injections (loading dose of 600mg subcutaneously followed by 300 mg subcutaneously every 2 weeks). One-third will receive placebo injections.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Active Comparator): Patients with severe hand eczema with an inadequate response or intolerance to alitretinoin. This group will receive dupilumab injections (600mg subcutaneously as a loading dose, followed by 300mg subcutaneously once every two weeks).
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Patients with severe hand eczema with an inadequate response or intolerance to alitretinoin. This group will receive placebo injections (600mg subcutaneously as a loading dose, followed by 300mg subcutaneously once every two weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab injections (blinded labels)
  Other Names: Dupixent
  Arms: Dupilumab
Drug: Placebo — Placebo injections (blinded labels), matching the dupilumab injections in quantity and appearance
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of dupilumab in hand eczema patients with an inadequate response or intolerance to alitretinoin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Severe or very severe chronic hand eczema as defined by a Physician Global Assessment (PGA) using a validated Photoguide.
* Inflammatory subtypes of hand eczema: recurrent vesicular hand eczema or chronic fissured hand eczema.
* An inadequate response to topical corticosteroids within 6 months before screening.
* A history of prior alitretinoin exposure and inadequate response or intolerance to alitretinoin.
* Patients has also received standard skin care, including emollients and barrier protection as appropriate, without significant improvement.
* Patients has avoided irritants and contact allergens, if identified, without significant improvement.
* Women of childbearing potential are required to use a highly effective (failure rate of <1% per year when used consistently and correctly) method of birth control, prior to receiving study intervention, during the study and for at least 10 weeks after receiving the last administration of study intervention. E.g., established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device or intrauterine system; barrier methods: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal foam/gel/film/cream/suppository (if available in their locale); male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant). NOTE: If a female participant's childbearing potential changes after start of the study (e.g., a woman who is not heterosexually active becomes active, a premenarchal woman experiences menarche), she must begin practicing a highly effective method of birth control, as described above.
* A woman of childbearing potential must have a negative serum or urine pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening and at Week 0 prior to administration of study intervention;
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 12 weeks after the last administration of study intervention.
* Agree not to receive a Bacillus Calmette-Guérin (BCG) vaccination during the study, or within 12 months after the last administration of study intervention.
* Be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, and is willing to participate in the study.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Other clinical subtypes of hand eczema, e.g. hyperkeratotic hand eczema, as defined by the Danish Contact Dermatitis Group24.
* Treatment with alitretinoin, systemic immunosuppressive medication or UV radiation within the previous 4 weeks.
* Patients with predominantly atopic dermatitis, in whom the hands are also involved, but no main concern. Patients with controlled atopic dermatitis, in which the hands are mainly affected, are eligible for inclusion.
* Psoriasis of the hands.
* Active bacterial, fungal, or viral infection of the hands.
* Pregnant/lactating or planning to become pregnant during the study period.
* Current malignancy (other than successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and⁄or localized carcinoma in situ of the cervix).
* Participant has known allergies, hypersensitivity, or intolerance to dupilumab or its excipients: L-arginine hydrochloride, L-histidine, polysorbate 80, sodium acetate, acetic acid, sucrose, water for injections.
* Participants with active helminth and other parasitic infections.
* Patients infected with human immunodeficiency virus (HIV) (positive serology for HIV antibody).
* Patients testing positive for hepatitis B virus (HBV) or hepatitis C (HCV) infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Response to treatment/hand eczema severity (Hand Eczema Severity Index, HECSI) | 16 weeks
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs of hand eczema and the extent of the lesions on each of 5 hand areas by use of standard scales. The total HECSI score is based on a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and a 5-point scale rating the affected area(s) ranging from 0 (0% affected area) to 4 (76% to 100% affected area). A decrease in score relates to an improvement in signs and symptoms. Response is defined as HECSI-75: the proportion of patients wit a HECSI score of ≥75% improvement from baseline.

SECONDARY OUTCOMES:
Response to treatment/hand eczema severity (Photographic guide) | Week 4, 8, 12, 16
  The photographic guide is a five-point scale that provides a global clinical assessment of hand eczema severity ranging from 0 to 4, where 0 indicates clear, 1 is almost clear, 2 is moderate, 4 is severe; and 5 indicates very severe hand eczema. A decrease in score relates to an improvement in signs and symptoms.
Response to treatment/hand eczema/foot eczema severity (Physician Global Assessment) | Week 4, 8, 12, 16
  A decrease in score relates to an improvement in signs and symptoms.
Response to treatment/hand eczema/foot eczema severity (modified Total Lesion Symptom Score, mTLSS) | Week 4, 8, 12, 16
  mTLSS combines an evaluation of hand and foot eczema lesions severity; scores are summed, extending from a base estimation of 0 (no signs or symptoms) to the most extreme of 18 (more serious disease).
Response to treatment/hand eczema severity (Hand Eczema Severity Index, HECSI) | Week 4, 8, 12, 16
  HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs of hand eczema and the extent of the lesions on each of 5 hand areas by use of standard scales. The total HECSI score is based on a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and a 5-point scale rating the affected area(s) ranging from 0 (0% affected area) to 4 (76% to 100% affected area). A decrease in score relates to an improvement in signs and symptoms.
Patient reported change (Patient Global Assessment, PaGA) | Week 4, 8, 12, 16
  Percentage of change of hand eczema symptoms assessed by PaGA. 0 indicates clear or almost clear (at least 90% clearing of disease signs and symptoms compared to baseline), 5 means worsening of symptoms compared to baseline.
Changeof pruritus (Numerical Rating Scale, NRS) | Week 4, 8, 12, 16
  Pruritus NRS is an assessment tool that is used to report the intensity of a patient's pruritus, both maximum and average intensity, during a 24-hour recall period. Maximum itch intensity on a scale of 0 - 10 (0 = no itch; 10 = worst itch imaginable).
Change of pain (Numerical Rating Scale, NRS) | Week 4, 8, 12, 16
  Pain NRS is an assessment tool that is used to report the intensity of a patient's pain, both maximum and average intensity, during a 24-hour recall period. Maximum pain intensity on a scale of 0 - 10 (0 = no pain; 10 = worst pain imaginable).
Change of hand eczema related quality of life (Quality of Life in Hand Eczema Questionnaire, QOLHEQ) | Week 4, 8, 12, 16
  The Quality Of Life in Hand Eczema Questionnaire (QOLHEQ) is an instrument to assess disease specific Health Related Quality of Life (HRQOL) in patients suffering from hand eczema. The construct HRQOL includes all impairments or limiting conditions caused by the health state of an individual. The QOLHEQ is a disease specific instrument, thereby only assessing impairments caused by hand eczema. It consists out of 30 items which can be summarized according to four domains of HRQOL: Impairments because of (1) symptoms, (2) emotions, (3) limitations in functioning or (4) because of treatment and prevention. A high score is indicative of a poor hand eczema related HRQOL.
Changeof quality of life (Dermatology Life Quality Index, DLQI) | Week 4, 8, 12, 16
  DLQI is a 10-item, validated questionnaire to assess the impact of skin disease symptoms and treatment on quality of life (QOL); over the past week, with an overall scoring of 0 (disease has no effect on patient's life) to 30 (disease has an extremely large effect on patient's life); a high score is indicative of a poor QoL.
Change of work productivity and impairment (Work Productivity and Activity Impairment, WPAI) | Week 4, 8, 12, 16
  The WPAI consists of 6 items, assessing absenteeism, presenteeism, work productivity loss and activity impairment. Higher scores indicate less productivity and a greater impairment.
Change of anxiety and depression (Hospital Anxiety and Depression scale, HADS) | Week 4, 8, 12, 16
  HADS is a 14-item questionnaire, 7 items for anxiety and 7 items for depression symptoms; possible scores range from 0 to 21 for each subscale. The following cut-off scores are recommended for both subscales: 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Cost-utility. Quality-adjusted life-years (QALY's): registered direct/indirect costs, combined with EQ-5D-5L outcome | Week 4, 8, 12, 16
Cost-effectiveness: registered direct/indirect costs combined with the primary and secondary effectiveness outcomes (HECSI and PG) | Week 4, 8, 12, 16
Safety and tolerability (adverse events) | Up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be published anonymously and will not be possible to trace back to individual participants.

REFERENCES:
- [Derived] Voorberg AN, Kamphuis E, Christoffers WA, Schuttelaar MLA. Efficacy and safety of dupilumab in patients with severe chronic hand eczema with inadequate response or intolerance to alitretinoin: a randomized, double-blind, placebo-controlled phase IIb proof-of-concept study. Br J Dermatol. 2023 Sep 15;189(4):400-409. doi: 10.1093/bjd/ljad156. PMID 37170922